CLINICAL TRIAL: NCT03592927
Title: Acute Exposure to Hypoxia in Precapillary Pulmonary Hypertension: Physiological and Clinical Effects at Rest and During Exercise
Brief Title: Acute Exposure to Simulated Hypoxia on Exercise Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-00455_A1
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Hypertension
Keywords: exercise capacity; simulated altitude
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Including a baseline assessment and assessments under simulated altitude and normoxia.
Who Masked: Participant
Masking Description: The allocated gas mixture will not be disclosed to the patient since he will breath through a facemask during both interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order A (Experimental): The participants will be exposed to shamed hypoxia (FiO2: 20.9% equivalent to sea level and consecutively to simulated altitude (FiO2: 15.1% equivalent to 2500m above sea level) administered by an altitude Simulator ("Altitrainer", SMTEC), simulated altitude (FiO2: 15.1%), with a facemask.
  Interventions: Device: Simulated Altitude (FiO2: 15.1%); Device: Shamed Hypoxia (FiO2: 20.9)
- Order B (Experimental): The participant will be exposed to hypoxia (FiO2, 15.1% equivalent to 2500m above sea level), simulated altitude (FiO2: 15.1%), and consecutively to shamed hypoxia (FiO2, 20.9%) administered by an altitude simulator ("Altitrainer", SMTEC) with a facemask.
  Interventions: Device: Simulated Altitude (FiO2: 15.1%); Device: Shamed Hypoxia (FiO2: 20.9)

INTERVENTIONS:
Device: Simulated Altitude (FiO2: 15.1%) — Inhalation of deoxygenated air through a altitude simulator ("Altitrainer"), for approx. 1 hour. given by a facemask.
Device: Shamed Hypoxia (FiO2: 20.9) — Inhalation of unmodified air through an altitude Simulator ("Altitrainer") for approximately 1 hour given by a facemask

SUMMARY:
Randomized crossover trial in patients with Pulmonary Hypertension (PAH, CTEPH) to assess the acute response to simulated altitude (FiO2:15.1, equivalent to 2500m above sea level) in constant loaded exercise capacity.

DETAILED DESCRIPTION:
Low altitude baseline measurements will be performed in Zurich (460m asl) including Echocardiography, Right heart catheterization, six-minute walk test (6MWT), pulmonary function test, clinical assessment and blood gas Analysis.

Randomly assigned to the order of testing, the participants will be tested under simulated altitude (FiO2: 15.1% with the "AMC Altitrainer") and shamed altitude with the same device.

Towards the end of the exposure after approximately 1h, the participants will perform a constant loaded exercise test on an Ergometer with a calculated resistance of their 60% max. workload.

The patients will be encouraged to perform this test up to their physical exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* PH diagnosed according to internation Guidelines: mean pulmonary artery presssure (mPAP) ≥ 25 mmHg along with a pulmonary artery wedge pressure (PAWP) ≤15 mmHg during right heart catheterization at the time of initial diagnosis
* PH class 1 (PAH) or 4 (CTEPH)
* Stable condition, on the same medication for > 4 weeks
* Patient live permanently at an altitude < 1000m asl.

Exclusion Criteria:

* Resting partial Oxygen pressure (PaO2) ≤7.3 kiloPascal (kPA) corresponding to the requirement of long-term oxygen therapy > 16hour daily (nocturnal oxygen therapy alone is allowed)
* Severe daytime hypercapnia (pCO2 > 6.5 kPa)
* Susceptibility to high altitude related diseases (AMS, High Altitude Pulmonary edema (HAPE), etc.) based on previous experienced discomfort at altitudes.
* Exposure to an altitude >1500m for ≥3 nights during the last 4 weeks before the study participation
* Residence > 1000m above sea level
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurological or orthopedic problems with walking disability
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Endurance time under hypoxia (FiO2: 15.1%) | Towards the end of a one hour exposure
  Constant loaded exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof., Principal Investigator — University of Zurich
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Schneider SR, Lichtblau M, Furian M, Mayer LC, Berlier C, Muller J, Saxer S, Schwarz EI, Bloch KE, Ulrich S. Cardiorespiratory Adaptation to Short-Term Exposure to Altitude vs. Normobaric Hypoxia in Patients with Pulmonary Hypertension. J Clin Med. 2022 May 14;11(10):2769. doi: 10.3390/jcm11102769. PMID 35628896
- [Derived] Schneider SR, Mayer LC, Lichtblau M, Berlier C, Schwarz EI, Saxer S, Furian M, Bloch KE, Ulrich S. Effect of Normobaric Hypoxia on Exercise Performance in Pulmonary Hypertension: Randomized Trial. Chest. 2021 Feb;159(2):757-771. doi: 10.1016/j.chest.2020.09.004. Epub 2020 Sep 9. PMID 32918899